CLINICAL TRIAL: NCT04824820
Title: Effect of Commercial Genital Vibrators Use on Female Wellness
Brief Title: Improving Female Sexual Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Karyn Eilber, Female Pelvic Medicine & Reconstructive Surgery Chair, Cedars-Sinai Medical Group Department of Surgery Associate Professor, Urology and Obstetrics & Gynecology, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00001138
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Sexuality; Sexual Dysfunction; Sexual Desire Disorder; Hypoactive Sexual Desire Disorder; Orgasmic Disorder; Pelvic Organ Prolapse; Urinary Incontinence; Interstitial Cystitis; Pelvic Floor Disorders; Female Sexual Dysfunction
Keywords: sexuality; Sexual Dysfunction; Sexual Desire Disorder; Hypoactive Sexual Desire Disorder; Orgasmic Disorder; Pelvic Organ Prolapse; Urinary Incontinence; Interstitial Cystitis; Pelvic Floor Disorders; Wellness; Female Sexual Dysfunction
MeSH Terms: conditions — Sexuality; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Pelvic Organ Prolapse; Urinary Incontinence; Cystitis, Interstitial; Pelvic Floor Disorders | interventions — Vib protein, Drosophila

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibrator (Experimental): Participants will be using commercially available genital vibrator for at least 5 minutes and/or reaching an orgasm three times a week for 3-4 months.
  Interventions: Behavioral: Vibrator

INTERVENTIONS:
Behavioral: Vibrator — Clitoral stimulation

SUMMARY:
The purpose of this study is to assess the effect of commercially available genital vibrator use on sexual health, female pelvic floor disorders, and overall quality of life among a diverse population of women.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Diagnosis of female sexual dysfunction, pelvic floor dysfunction, genito-urologic issues (stress urinary incontinence, urge urinary incontinence, pelvic organ prolapse, interstitial cystitis, pelvic pain, dyspareunia, lichen sclerosis)
* Manual dexterity to use vibrator

Exclusion Criteria:

* Non English speaking
* Pregnancy or <12 months postpartum
* Poor manual dexterity

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
To assess the change from baseline sexual function at 3 month | baseline, post intervention at 3 months
  Assessment based on validated questionnaire. Female Sexual Function Index (FSFI), a 19-item measure of sexual function in all four domains: desire, arousal, orgasm and sexual pain. The total score ranges from 0-36, with higher scores indicating better sexual function. Total score below 26.6 indicates clinical Female Sexual Dysfunction (FSD).
To assess the change from baseline sexual function at 3 month | baseline, post intervention at 3 months
  Assessment based on validated questionnaire. The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire International Urogynecological Association (IUGA) Revised (PISQ-IR) is a validated measure of sexual function among not only sexually active women but also sexually inactive women. This questionnaire contains 20 questions, and is used to assess sexual activity in women with urinary incontinence and pelvic organ prolapse. The higher the score the better the Sexual Function.
To assess the change from baseline degree of pelvic organ prolapse at 3 month | baseline, post intervention at 3 months
  The Pelvic Organ Prolapse Quantifications System (POP-Q) is a system for assessing the degree of prolapse of pelvic organs to help standardize diagnosing, comparing, documenting, and sharing of clinical findings. This assessment is the most frequently used among research publications related to pelvic organ prolapse.
To assess the change from baseline overall health and quality of life at 3 month | baseline, post intervention at 3 months
  Self-reported quality of life (SF-12) is a general health measure assessing the impact of health on an individual's everyday life. The SF-12 consists of eight domains and generates two separate summary scores, physical functional scores (PCS) and mental function scores (MCS), ranging from 0 to 100. Higher scores indicated better health related quality of life.
To assess the change from baseline overall health and quality of life at 3 month | baseline, post intervention at 3 months
  Patient Health Questionnaire (PHQ-9) is a tool to assess depression. The severity of depression is assessed by summarizing the scores assigned to the categories, with score ranging between 1 and 27, with higher score correlating with more sever depression.
To assess the change from baseline overall health and quality of life at 3 month | baseline, post intervention at 3 months
  The Pelvic Floor Distress Inventory Questionnaire (PFDI) is a condition-specific quality-of-life questionnaire for women with bowel, bladder, and/or pelvic symptoms. The scores range between 0 to 300 with higher scores indicating more severe distress.

CONTACTS AND LOCATIONS:
Overall Officials: Karyn Eilber, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No